CLINICAL TRIAL: NCT07290127
Title: Effects of a Computer Game on Postpartum Mental Health After Emergency Cesarean Birth: a Feasibility Randomized Controlled Trial
Brief Title: A Computer Game for Postpartum Mental Health After Emergency Cesarean Birth
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kyoto University, Graduate School of Medicine (Other)
Responsible Party: Principal Investigator, Sachiko Asada, Principal Investigator, Kyoto University, Graduate School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C1606
Record Dates: First submitted 2025-06-30; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Post-traumatic Stress Disorder (PTSD); Postpartum Mental Health
Keywords: post-traumatic stress disorder; PTSD; postpartum; mental health; emergency caesarean birth; randomised controlled trial; computer game; Tetris; pilot study; feasibility study
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: implementation of a brief computer-based intervention "Tetris"
- Usual care group (No Intervention)

INTERVENTIONS:
Behavioral: implementation of a brief computer-based intervention "Tetris" — Within 24 hours of emergency caesarean birth, the participants played Tetris (TetrisⓇ99), a cognitive task, for at least 10 and up to 15 minutes on a Nintendo Switch Lite game console.
  Arms: Intervention group

SUMMARY:
This study aims to explore whether playing the computer game Tetris can reduce PTSD symptoms in women who have undergone emergency caesarean births. Additionally, as a feasibility study, it seeks to provide essential data and insights that will guide the design and implementation of future larger-scale RCTs examining the effects of Tetris in this context.

The specific objectives are to explore:

1. Whether playing Tetris within 24 hours of an emergency C-section help to reduce symptoms of PTSD.
2. Clinical feasibility and acceptability for an intervention (ie. game Tetris) immediately after a cesarean section.
3. Issues arising from the research design, including requitement and sample size.

Participants in the intervention group will play Tetris for at least 10 minutes, but no more than 15 minutes within 24 hours of a C-section.

For outcomes, all participants will complete the questionnaires on the fifth day after the C-section and one month postpartum.

DETAILED DESCRIPTION:
Recent research suggests that adverse events related to childbirth and pregnancy, such as emergency caesarean births, can trigger post-traumatic stress disorder (PTSD). Although therapeutic and preventive interventions like trauma-focused cognitive behavioural therapy (CBT) are available, the effectiveness of interventions that do not require specialist expertise remains unclear.

This randomised controlled trial (RCT) aims to determine whether playing the computer game Tetris can reduce the PTSD symptom severity in postpartum women who have undergone emergency caesarean births, a group at higher risk of developing PTSD compared to those who have had spontaneous deliveries. Additionally, this study serves as a feasibility test, establishing a foundation for future larger RCTs examining the effects of Tetris.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20 years or older
* Women who have undergone an emergency caesarean birth within the previous 24 hours
* Must be able to understand instructions and respond to the questionnaire in Japanese

Exclusion Criteria:

* Undergoing treatment for psychiatric disorders such as PTSD, depression, anxiety disorders or schizophrenia.
* Undergoing intensive care after surgery .
* The physician does not approve participation for any physical or mental reasons .

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2025-12-13 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Impact of Event Scale-Revised (IES-R) scores (intrusive, avoidance and total scores) at one month postpartum | At one month postpartum
  The participants are asked to report the degree of distress experienced for each item in the past 7 days. The 5 points on the scale are: 0 (not at all), 1 (a little bit), 2 (moderately), 3 (quite a bit), 4 = (extremely).

SECONDARY OUTCOMES:
IES-R at 5 days postpartum | At 5 days postpartum
  The participants are asked to report the degree of distress experienced for each item in the past 7 days. The 5 points on the scale are: 0 (not at all), 1 (a little bit), 2 (moderately), 3 (quite a bit), 4 = (extremely).
Edinburgh Postnatal Depression Scale (EPDS) at 5 days and one month postpartum | At 5 days and one month postpartum
  Each of the 10 questions has four possible responses, with scores ranging from 0 to 3. The scores for all 10 items are then added together to get a total score.
Labour Agentry Scale (LAS) at 5 days and one month postpartum | At 5 days and one month postpartum
  The LAS is a 29-item scale with a single underlying factor relating to mastery and sense of control. It has high internal reliability. The scale includes a 10-item inventory with six positive and four negative descriptions of the perceived degree of control experienced during childbirth. Participants ranked the items on a seven-point scale ranging from (1) "almost all of the time" to (7) "never, or almost never."
Social Support Questionnaire (SSQ) at 5 days and one month postpartum | At 5 days and one month postpartum
  The SSQ is a 6-item questionnaire designed to measure perceptions of and satisfaction with social support. Each item is a question that solicits a two-part answer. The first part asks participants to list all the people that fit the description of the question. The SSQ number score is calculated by adding the total number of responses to all six questions (with a minimum of 0 and no maximum) and dividing by 6 to find the average item score. The second part asks participants to indicate how satisfied they are, in general, with these people. The SSQ satisfaction score is calculated by adding the total number of responses to all six questions (with a minimum of 6 to a maximum of 36) and dividing by six to find the average item score.
Breastfeeding Status | At 5 days and one month postpartum
  Type of nutritional method of the newborn .
Number of medical visits and consultations | At one month postpartum
  Number of visits to medical institutions and telephone consultations after discharge at the 1-month checkup.

OTHER OUTCOMES:
The number of women who met the eligibility criteria but declined to participate in the study and their reasons for doing so. | At one month postpartum
  Feasibility of computer game intervention in the intervention group. The range is from 0 to no upper limit.
Follow-up rate | At one month postpartum
  Percentage of participants who were followed from the beginning of the study until one month postpartum. The range is from 0% to 100%.
Questionnaire response rate. | At one month postpartum.
  Percentage of respondents who answered all the questions. The range is from 0% to 100%.
Adherence/compliance rate. | Within 24 hours after a cesarean section.
  Percentage of intervention group participants who correctly played computer games for the specified amount of time. The range is from 0% to 100%.
Reasons for dropping out. | Within 24 hours after a cesarean section, at 5 days and one month postpartum.
  Describe the reasons why participants dropped out of the study during the research process to evaluate its feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Sachiko Asada, Master's degree, Principal Investigator — Perinatal epidemiology Department of Human Health Sciences Graduate School of Medicine Kyoto University; Marie Furuta, Ph.D., Study Chair — Perinatal epidemiology Department of Human Health Sciences Graduate School of Medicine Kyoto University
Locations (1):
- Perinatal epidemiology Department of Human Health Sciences Graduate School of Medicine Kyoto University, Kyoto, Sakyo-ku, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Paul IM, Downs DS, Schaefer EW, Beiler JS, Weisman CS. Postpartum anxiety and maternal-infant health outcomes. Pediatrics. 2013 Apr;131(4):e1218-24. doi: 10.1542/peds.2012-2147. Epub 2013 Mar 4. PMID 23460682
- [Result] Turkstra E, Creedy DK, Fenwick J, Buist A, Scuffham PA, Gamble J. Health services utilization of women following a traumatic birth. Arch Womens Ment Health. 2015 Dec;18(6):829-32. doi: 10.1007/s00737-014-0495-7. Epub 2015 Jan 11. PMID 25577338
- [Result] Dias CC, Figueiredo B. Breastfeeding and depression: a systematic review of the literature. J Affect Disord. 2015 Jan 15;171:142-54. doi: 10.1016/j.jad.2014.09.022. Epub 2014 Sep 28. PMID 25305429
- [Result] Cook N, Ayers S, Horsch A. Maternal posttraumatic stress disorder during the perinatal period and child outcomes: A systematic review. J Affect Disord. 2018 Jan 1;225:18-31. doi: 10.1016/j.jad.2017.07.045. Epub 2017 Jul 27. PMID 28777972
- [Result] World Health Organization(2008）: Indicators for assessing infant and young child feeding practices : conclusions of a consensus meeting held 6-8 November 2007 in Washington D.C. ,USA.
- [Result] Furukawa TA, Harai H, Hirai T, Kitamura T, Takahashi K. Social Support Questionnaire among psychiatric patients with various diagnoses and normal controls. Soc Psychiatry Psychiatr Epidemiol. 1999 Apr;34(4):216-22. doi: 10.1007/s001270050136. PMID 10365628
- [Result] Sarason IG, Levine HM, Basham RB, Sarason BR(1983): Assessing Social Support: The Social Support Questionnaire. Journal of Personality and Social Psychology 44(1)127-139.
- [Result] Gurber S, Baumeler L, Grob A, Surbek D, Stadlmayr W. Antenatal depressive symptoms and subjective birth experience in association with postpartum depressive symptoms and acute stress reaction in mothers and fathers: A longitudinal path analysis. Eur J Obstet Gynecol Reprod Biol. 2017 Aug;215:68-74. doi: 10.1016/j.ejogrb.2017.05.021. Epub 2017 May 30. PMID 28601730
- [Result] 毛利多恵子（1994）：産婦の身体拘束が陣痛体験に及ぼす影響．1993年度聖路加看護大学大学院修士論文
- [Result] Hodnett ED, Simmons-Tropea DA. The Labour Agentry Scale: psychometric properties of an instrument measuring control during childbirth. Res Nurs Health. 1987 Oct;10(5):301-10. doi: 10.1002/nur.4770100503. PMID 3671777
- [Result] 岡野 禎, 村田 真, 増地 聡, 他（1996） 日本版エジンバラ産後うつ病自己評価票(EPDS)の信頼性と妥当性. 精神科診断学. 7(4):525-533.
- [Result] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Result] Asukai N, Kato H, Kawamura N, Kim Y, Yamamoto K, Kishimoto J, Miyake Y, Nishizono-Maher A. Reliability and validity of the Japanese-language version of the impact of event scale-revised (IES-R-J): four studies of different traumatic events. J Nerv Ment Dis. 2002 Mar;190(3):175-82. doi: 10.1097/00005053-200203000-00006. PMID 11923652
- [Result] Weiss DS(2004): The Impact of Event Scale-Revised. In: Wilson, J.P., Keane T.M. eds., Assessing psychological trauma and PTSD（Second Edition）. The Guilford Press, New York, 168-189.
- [Result] Ayers S, Rados SN, Balouch S. Narratives of traumatic birth: Quality and changes over time. Psychol Trauma. 2015 May;7(3):234-42. doi: 10.1037/a0039044. PMID 25961868
- [Result] Adshead G. Psychological therapies for post-traumatic stress disorder. Br J Psychiatry. 2000 Aug;177:144-8. doi: 10.1192/bjp.177.2.144. PMID 11026954
- [Result] Horsch A, Vial Y, Favrod C, Harari MM, Blackwell SE, Watson P, Iyadurai L, Bonsall MB, Holmes EA. Reducing intrusive traumatic memories after emergency caesarean section: A proof-of-principle randomized controlled study. Behav Res Ther. 2017 Jul;94:36-47. doi: 10.1016/j.brat.2017.03.018. Epub 2017 Apr 6. PMID 28453969
- [Result] Monfils MH, Cowansage KK, Klann E, LeDoux JE. Extinction-reconsolidation boundaries: key to persistent attenuation of fear memories. Science. 2009 May 15;324(5929):951-5. doi: 10.1126/science.1167975. Epub 2009 Apr 2. PMID 19342552
- [Result] Krans J, Naring G, Holmes EA, Becker ES. Motion effects on intrusion development. J Trauma Dissociation. 2010;11(1):73-82. doi: 10.1080/15299730903318483. PMID 20063249
- [Result] Lilley SA, Andrade J, Turpin G, Sabin-Farrell R, Holmes EA. Visuospatial working memory interference with recollections of trauma. Br J Clin Psychol. 2009 Sep;48(Pt 3):309-21. doi: 10.1348/014466508X398943. Epub 2009 Jan 30. PMID 19187579
- [Result] James EL, Bonsall MB, Hoppitt L, Tunbridge EM, Geddes JR, Milton AL, Holmes EA. Computer Game Play Reduces Intrusive Memories of Experimental Trauma via Reconsolidation-Update Mechanisms. Psychol Sci. 2015 Aug;26(8):1201-15. doi: 10.1177/0956797615583071. Epub 2015 Jul 1. PMID 26133572
- [Result] Kida S. Reconsolidation/destabilization, extinction and forgetting of fear memory as therapeutic targets for PTSD. Psychopharmacology (Berl). 2019 Jan;236(1):49-57. doi: 10.1007/s00213-018-5086-2. Epub 2018 Oct 29. PMID 30374892
- [Result] Abel T, Lattal KM. Molecular mechanisms of memory acquisition, consolidation and retrieval. Curr Opin Neurobiol. 2001 Apr;11(2):180-7. doi: 10.1016/s0959-4388(00)00194-x. PMID 11301237
- [Result] McGaugh JL. Memory--a century of consolidation. Science. 2000 Jan 14;287(5451):248-51. doi: 10.1126/science.287.5451.248. PMID 10634773
- [Result] Gentile M a,b, Lieto A(2022): The role of mental rotation in TetrisTM gameplay: An ACT-R computational cognitive model. Cognitive Systems Research 73 1-11.
- [Result] Walker MP, Brakefield T, Hobson JA, Stickgold R. Dissociable stages of human memory consolidation and reconsolidation. Nature. 2003 Oct 9;425(6958):616-20. doi: 10.1038/nature01930. PMID 14534587
- [Result] Brewin CR. Episodic memory, perceptual memory, and their interaction: foundations for a theory of posttraumatic stress disorder. Psychol Bull. 2014 Jan;140(1):69-97. doi: 10.1037/a0033722. Epub 2013 Aug 5. PMID 23914721
- [Result] Astill Wright L, Horstmann L, Holmes EA, Bisson JI. Consolidation/reconsolidation therapies for the prevention and treatment of PTSD and re-experiencing: a systematic review and meta-analysis. Transl Psychiatry. 2021 Sep 3;11(1):453. doi: 10.1038/s41398-021-01570-w. PMID 34480016
- [Result] Iyadurai L, Blackwell SE, Meiser-Stedman R, Watson PC, Bonsall MB, Geddes JR, Nobre AC, Holmes EA. Preventing intrusive memories after trauma via a brief intervention involving Tetris computer game play in the emergency department: a proof-of-concept randomized controlled trial. Mol Psychiatry. 2018 Mar;23(3):674-682. doi: 10.1038/mp.2017.23. Epub 2017 Mar 28. PMID 28348380
- [Result] Kanstrup M, Singh L, Goransson KE, Widoff J, Taylor RS, Gamble B, Iyadurai L, Moulds ML, Holmes EA. Reducing intrusive memories after trauma via a brief cognitive task intervention in the hospital emergency department: an exploratory pilot randomised controlled trial. Transl Psychiatry. 2021 Jan 11;11(1):30. doi: 10.1038/s41398-020-01124-6. PMID 33431807
- [Result] Slade PP, Molyneux DR, Watt DA. A systematic review of clinical effectiveness of psychological interventions to reduce post traumatic stress symptoms following childbirth and a meta-synthesis of facilitators and barriers to uptake of psychological care. J Affect Disord. 2021 Feb 15;281:678-694. doi: 10.1016/j.jad.2020.11.092. Epub 2020 Nov 11. PMID 33220947
- [Result] de Graaff LF, Honig A, van Pampus MG, Stramrood CAI. Preventing post-traumatic stress disorder following childbirth and traumatic birth experiences: a systematic review. Acta Obstet Gynecol Scand. 2018 Jun;97(6):648-656. doi: 10.1111/aogs.13291. Epub 2018 Mar 2. PMID 29336486
- [Result] Furuta M, Horsch A, Ng ESW, Bick D, Spain D, Sin J. Effectiveness of Trauma-Focused Psychological Therapies for Treating Post-traumatic Stress Disorder Symptoms in Women Following Childbirth: A Systematic Review and Meta-Analysis. Front Psychiatry. 2018 Nov 20;9:591. doi: 10.3389/fpsyt.2018.00591. eCollection 2018. PMID 30515108
- [Result] Takeda S, Takeda J, Murakami K, Kubo T, Hamada H, Murakami M, Makino S, Itoh H, Ohba T, Naruse K, Tanaka H, Kanayama N, Matsubara S, Sameshima H, Ikeda T. Annual Report of the Perinatology Committee, Japan Society of Obstetrics and Gynecology, 2015: Proposal of urgent measures to reduce maternal deaths. J Obstet Gynaecol Res. 2017 Jan;43(1):5-7. doi: 10.1111/jog.13184. PMID 28074548
- [Result] Gradus JL, Qin P, Lincoln AK, Miller M, Lawler E, Sorensen HT, Lash TL. Posttraumatic stress disorder and completed suicide. Am J Epidemiol. 2010 Mar 15;171(6):721-7. doi: 10.1093/aje/kwp456. Epub 2010 Feb 16. PMID 20160171
- [Result] Yildiz PD, Ayers S, Phillips L. The prevalence of posttraumatic stress disorder in pregnancy and after birth: A systematic review and meta-analysis. J Affect Disord. 2017 Jan 15;208:634-645. doi: 10.1016/j.jad.2016.10.009. Epub 2016 Oct 27. PMID 27865585
- [Result] Grisbrook MA, Dewey D, Cuthbert C, McDonald S, Ntanda H, Giesbrecht GF, Letourneau N. Associations among Caesarean Section Birth, Post-Traumatic Stress, and Postpartum Depression Symptoms. Int J Environ Res Public Health. 2022 Apr 18;19(8):4900. doi: 10.3390/ijerph19084900. PMID 35457767
- [Result] Carter J, Bick D, Gallacher D, Chang YS. Mode of birth and development of maternal postnatal post-traumatic stress disorder: A mixed-methods systematic review and meta-analysis. Birth. 2022 Dec;49(4):616-627. doi: 10.1111/birt.12649. Epub 2022 May 13. PMID 35561055
- [Result] Williams C, Patricia Taylor E, Schwannauer M. A WEB-BASED SURVEY OF MOTHER-INFANT BOND, ATTACHMENT EXPERIENCES, AND METACOGNITION IN POSTTRAUMATIC STRESS FOLLOWING CHILDBIRTH. Infant Ment Health J. 2016 May;37(3):259-73. doi: 10.1002/imhj.21564. Epub 2016 Apr 19. PMID 27090507
- [Result] Ayers S, Bond R, Bertullies S, Wijma K. The aetiology of post-traumatic stress following childbirth: a meta-analysis and theoretical framework. Psychol Med. 2016 Apr;46(6):1121-34. doi: 10.1017/S0033291715002706. Epub 2016 Feb 16. PMID 26878223
- [Result] Dekel S, Stuebe C, Dishy G. Childbirth Induced Posttraumatic Stress Syndrome: A Systematic Review of Prevalence and Risk Factors. Front Psychol. 2017 Apr 11;8:560. doi: 10.3389/fpsyg.2017.00560. eCollection 2017. PMID 28443054
- [Result] Howard LM, Molyneaux E, Dennis CL, Rochat T, Stein A, Milgrom J. Non-psychotic mental disorders in the perinatal period. Lancet. 2014 Nov 15;384(9956):1775-88. doi: 10.1016/S0140-6736(14)61276-9. Epub 2014 Nov 14. PMID 25455248